CLINICAL TRIAL: NCT05525169
Title: Study of the Impact of Exposure to Outdoor and Indoor Pollutants in Patients With Asthma
Acronym: EXAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0115
Record Dates: First submitted 2022-07-07; First posted 2022-09-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Asthma
Keywords: Asthma; exacerbations; outdoor and indoor air pollutants
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project is to measure exposure to outdoor and indoor air pollutants in asthma patients in order to show a possible association between variation in pollutant exposure and the occurrence of exacerbations in these patients

DETAILED DESCRIPTION:
Asthma is a chronic airway disease affecting between 6% and 7% of the French adult population. Asthma is responsible for nearly 1000 deaths each year in France. Air pollution (indoor and outdoor) is responsible for 7 million deaths each year according to the World Health Organization (WHO) assessment published in 2018, including 65,000 in France. Studies monitoring exposure to indoor air pollutants are few in number in asthmatic patients. Very little research has been devoted to continuous monitoring of indoor air quality in homes. Our hypothesis is that variation in exposure to indoor air pollutants, in relation to outdoor air, would have an impact on the occurrence of exacerbations in asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* Patient with a confirmed diagnosis of asthma for at least 12 months as defined by the investigator,
* Patient with at least 4 asthma exacerbations in the last year
* Patient sleeping at least 6 nights per week in the same home

Exclusion Criteria:

* Patient who is an active smoker or living with an active smoker,
* Patient with a diagnosis of COPD, ABPA or associated pulmonary fibrosis,
* Patient with an asthma exacerbation within 15 days prior to the inclusion visit,
* Patient with known occupational exposure,
* Patient living in a dwelling that does not allow the installation of sensors (inability to connect the sensor to the power supply, no location for the outdoor sensor...)
* Patient who plans to move in the next 6 months,
* Patient with a life expectancy of less than 6 months,
* Patient who has someone living in their household also included in EXAP,
* Patient who lives in an apartment and does not have a balcony or space for the outdoor sensor,
* Pregnant or breastfeeding women,

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult men and women recruited from the active file of asthma patients followed at the Nantes University Hospital, the Saint Nazaire Hospital, the Châteaubriant Nozay Pouancé Hospital and the Erdre et Loire Hospital. Regardless of the type of asthma, patients will be potentially included if they have a minimum of 4 exacerbations during the year preceding inclusion in the EXAP project>. Participation in other non-interventional research is allowed during the study unless this research increases the number of exacerbations.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Asthma exacerbations | 36 months
  The primary criterion is the association between the occurrence of exacerbations and the concentrations of the following pollutants or other environmental factors measured daily in the patients' homes by air pollution sensor inside and outside the home.
  * the concentration of indoor pollutants: PM1 (µg/m3), PM2.5 (µg/m3), PM10 (µg/m3), volatile organic compounds (VOC) (µg/m3) , CO2 (ppm),
  * the concentration of outdoor pollutants (µg/m3): PM1, PM2.5, PM10,
  * The ratios (indoor/outdoor air) of PM1, PM2.5 and PM10 in the home,
  * Temperature(°C) and relative humidity (RH) (%) in indoor and outdoor air,
  * Exceedances of regulatory (provided by the Environmental Code) or recommended (determined by the sensor supplier) pollutant thresholds.

SECONDARY OUTCOMES:
Daily Peak flow (l/ min) | 36 months
  The secondary criterion is the the temporal association between the daily Peak flow and the concentrations of the same pollutants or other environmental factors listed in the primary criterion.
  Subgroup analyses : groups of patients will be created according to the characteristics of their habitat (heating mode, ventilation, rural or urban area...).
  Both primary and secondary outcomes will be studied in these subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier Blanc, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France